CLINICAL TRIAL: NCT05800626
Title: Prediction of Post-Endoscopic Retrograde Cholangio-Pancreatography Pancreatitis Based on the Appearance of the Major Duodenal Papilla: a Prospective, Observational, Cohort Study
Brief Title: Prediction of PEP Based on the Appearance of the Major Duodenal Papilla
Acronym: PredERCP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5534
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-03

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangio-Pancreatography (ERCP) — ERCP performed for clinical practice

SUMMARY:
This observational, prospective study aims at evaluating how the occurrence of post-Endoscopic Retrograde CholangioPancreatography (ERCP) acute pancreatitis (PEP) could be influenced by difficult biliary cannulation that might be previously assessed by the morphological appearance of native major papilla in all the patients undergoing ERCP.

The rate of successful biliary cannulation across papilla types could be used as intraprocedural quality and competence metrics during training. Moreover, recognizing difficult papillae could allow reserving those to experts to decrease the odds of failed cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with native duodenal papilla;
* Any indication to ERCP +/- biliary sphincterotomy of duodenal major papilla;
* Patients able to provide a written informed consent

Exclusion Criteria:

* ERCP performed for disorders unrelated to biliary tract;
* Previous upper gastrointestinal tract surgery;
* Presence of a duodenal stricture (either malignant or benign);
* Presence of a malignant infiltration of the papilla;
* Concomitant anticoagulant and/or P2Y12 inhibitors therapy (clopidogrel, prasugrel, ticagrelor) that precludes the treatment;
* INR > 1.5;
* Platelets count < 80000/mm3;
* Unwillingness to sign written informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all consecutive patients with a native major duodenal papilla undergoing ERCP. Patients that previously underwent ERCP with sphincterotomy will not be included. Patients will be considered enrolled after signing the informed consent form. All patients will be hospitalized for at least 24 hours after ERCP for clinical observation.
Sampling Method: Probability Sample
Enrollment: 1740 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of PEP occurrence | within 48 hours after the procedure
  Rate of PEP occurrence distributed between the different native major duodenal papilla types

SECONDARY OUTCOMES:
Rate of difficult biliary cannulation | during the procedure
  Rate of difficult biliary cannulation (> 5 cannulation attempts and/or > 5 minutes attempting to cannulate biliary duct and/or at least one passage in the pancreatic duct) distributed between the different native major duodenal papilla types
Rate of difficult biliary cannulation | during the procedure
  Rate of difficult biliary cannulation distributed between the different types of the intramural papillary segments on fluoroscopic images
Rate of intraoperative complications | during the procedure
  Rate of intraoperative complications distributed between the different native major duodenal papilla types
Rate of postoperative complications except for PEP | within 48 hours after the procedure
  Rate of postoperative complications except for PEP (up to 48 hours after ERCP) distributed between the different native major duodenal papilla types
Difference in the rate of difficult biliary cannulation | during the procedure
  Difference in the rate of difficult biliary cannulation between ERCP experts (>300 performed procedures) and fellows (<300 performed procedures)
occurrence of intra- and post-procedural complications | within 48 hours after the procedure
  To evaluate the occurrence of intra- and post-procedural complications but PEP, fluoroscopic morphology of the papillary segment of distal bile duct, perioperative and intraoperative risk factors

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma